CLINICAL TRIAL: NCT00072345
Title: A Phase II Study of Temozolomide, Thalidomide, and Lomustine in the Treatment of Advanced Melanoma
Brief Title: Temozolomide, Thalidomide, and Lomustine in Treating Patients With Unresectable Stage III or Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 03-084; P30CA008748 (NIH); MSKCC-03084
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Intraocular Melanoma; Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma; recurrent melanoma; iris melanoma; ciliary body and choroid melanoma, medium/large size; ciliary body and choroid melanoma, small size; extraocular extension melanoma; recurrent intraocular melanoma
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — Lomustine; Temozolomide; Thalidomide

INTERVENTIONS:
Drug: lomustine
Drug: temozolomide
Drug: thalidomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide and lomustine, use different ways to stop tumor cells from dividing so they stop growing or die. Thalidomide may stop the growth of cancer by stopping blood flow to the tumor. Combining temozolomide and thalidomide with lomustine may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining temozolomide and thalidomide with lomustine in treating patients who have unresectable stage III or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the antitumor activity of temozolomide, thalidomide, and lomustine, in terms of objective response rate, in patients with unresectable stage III or stage IV melanoma.

Secondary

* Determine the toxicity profile of this regimen in these patients.
* Determine the duration of response and overall survival of patients treated with this regimen.

OUTLINE: Patients receive oral temozolomide on days 1-42, oral thalidomide on days 1-56, and oral lomustine on days 1 and 29. Courses repeat every 8 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 12-35 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic malignant melanoma

  * Unresectable stage III OR stage IV disease
  * Ocular, mucosal, and cutaneous melanoma allowed
* Measurable disease

  * Indicator lesions within a prior radiotherapy field must have recent evidence of disease progression
  * Indicator lesions must be distinct from the surgical and/or radiation changes induced by prior local therapies
* No more than 2 symptomatic hemorrhagic lesions in the brain

  * No hemorrhagic lesion(s) greater than 1 cm in diameter

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 80-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* SGOT and SGPT no greater than 2 times ULN
* Alkaline phosphatase no greater than 2 times ULN
* Lactic dehydrogenase no greater than 2 times ULN

Renal

* Creatinine no greater than 2 mg/dL

Cardiovascular

* No history of severe cardiovascular disease
* No myocardial infarction within the past 6 months
* No unstable angina
* No New York Heart Association class III or IV congestive heart failure
* No ventricular arrhythmia
* No uncontrolled arrhythmia

Gastrointestinal

* No frequent vomiting
* No other medical condition that would preclude oral medication intake (e.g., partial bowel obstruction)

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 4 weeks after study participation
* HIV negative
* No AIDS-related illness
* No serious infection requiring IV antibiotics
* No other uncontrolled medical illness that would preclude study participation
* No other malignancy within the past 2 years except nonmelanoma skin cancer, carcinoma in situ of the cervix, or T1a or b prostate cancer meeting all of the following criteria:

  * Detected incidentally at transurethral resection of the prostate (TURP)
  * Comprises less than 5% of resected tissue
  * Prostate-specific antigen normal since TURP

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 3 weeks since prior immunotherapy or biologic therapy
* No concurrent immunotherapy

Chemotherapy

* No prior systemic chemotherapy for melanoma
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* At least 3 weeks since prior focused radiotherapy for brain metastases
* At least 3 weeks since prior radiosurgery
* At least 4 weeks since prior whole brain radiotherapy
* At least 3 weeks since prior interstitial brachytherapy
* No concurrent radiotherapy

Surgery

* See Disease Characteristics
* At least 3 weeks since prior surgery for brain metastases
* At least 3 weeks since prior surgery requiring general anesthesia

Other

* Recovered from all prior therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-07; Primary Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Jen Hwu, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States